CLINICAL TRIAL: NCT01293981
Title: Radiographic and Clinical Outcomes of PureGen Osteoprogenitor Cell Allograft in Posterior Lumbar and Transforaminal Interbody Fusion Procedures
Brief Title: Radiographic and Clinical Outcomes of PureGen in Posterior Lumbar (PLIF) and Transforaminal Interbody Fusion (TLIF)
Status: Terminated | Type: Observational
Why Stopped: Product no longer on the market
Sponsor: Alphatec Spine, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO-000058
Record Dates: First submitted 2011-02-09; First posted 2011-02-11 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Lumbar Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Lumbar Degenerative Disc Disease
  Interventions: Biological: PureGen Osteoprogenitor Cell Allograft

INTERVENTIONS:
Biological: PureGen Osteoprogenitor Cell Allograft — PureGen Osteoprogenitor Cell Allograft.

SUMMARY:
The purpose of this study is to assess the safety and efficacy of PureGen Osteoprogenitor Cell Allograft in patients undergoing Posterior Lumbar or Transforaminal Interbody Fusion.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with back and/or leg pain electing to receive Transforaminal Lumbar Interbody Fusion (TLIF)/ Posterior Lumbar Interbody Fusion (PLIF) procedure and posterior transpedicular stabilization with or without decompression at any level
* Unresponsive to conservative treatment for at least 6 months
* Radiographic confirmation of primary diagnosis

Exclusion Criteria:

* More than 2 levels requiring lumbar interbody fusion
* Spondylolisthesis greater than Grade I
* Prior failed fusion surgery at any lumbar level(s)
* Local or systemic infection past or present
* Active systemic disease
* Osteoporosis, osteomalacia, or other metabolic bone disease that would significantly inhibit bone healing
* BMI greater than 40
* Use of other bone graft, Bone Morphogenetic Protein (BMP) or bone graft substitutes in addition to or in place of those products specified
* Use of post operative Spinal Cord Stimulator (SCS)
* Any condition requiring postoperative medications that inhibit fusion, such as chronic use of oral or injected steroids or prolonged use of non-steroidal anti-inflammatory drugs
* Known or suspected history of alcohol and/or drug abuse
* Involved in pending litigation or worker's compensation related to the spine
* Pregnant or plans to become pregnant during the course of the study
* Insulin-dependent diabetes mellitus
* Known sensitivity to device materials
* Life expectancy less than duration of study
* Any significant psychological disturbance that could impair consent process or ability to complete self-assessment questionnaires
* Undergoing chemotherapy or radiation treatment
* Known history of hypersensitivity or anaphylactic reaction to dimethyl sulfoxide (DMSO)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects diagnosed with symptomatic lumbar degenerative disc disease (DDD) at 1 or 2 contiguous levels between L1 and S1.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2011-02; Primary Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Fusion | 24 months
  Proportion of subjects with fusion at the 24 month visit

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Beverly Hills, California
  - Middleton, Connecticut
  - Greensboro, North Carolina